CLINICAL TRIAL: NCT05538351
Title: A Study to Support the Development of the Enhanced Fluid Assessment Tool for Patients With Acute Kidney Injury
Status: Active, not recruiting | Type: Observational
Sponsor: University of Hertfordshire (Other)
Collaborators: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: HSK/PGR/NHS/02973
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: dehydration; hypotension; Acute Kidney Injury; hypovolaemia; respiratory rate; extracellular fluid; hypertension; body weight changes; pulmonary oedema; oedema; signs and symptoms; blood volume
MeSH Terms: conditions — Acute Kidney Injury; Dehydration; Hypotension; Hypovolemia; Hypertension; Body Weight Changes; Pulmonary Edema; Edema; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fluid assessment: All patients enrolled in this study will have a clinical assessment to identify hydration status, patient reported signs and symptoms of hydration and Bioimpedance using the Body composition Monitor (BCM).
  Interventions: Device: Body Composition Monitor (BCM)

INTERVENTIONS:
Device: Body Composition Monitor (BCM) — The hydration status of each participant from the clinical assessment and the patient reported signs and symptoms will be compared with the readings from bioimpedance (BCM machine).
  Other Names: Bioimpedance

SUMMARY:
Acute Kidney Injury (AKI) is the sudden and recent reduction in kidney function. This can be detected by measuring a rise in blood creatinine level or from a reduction in urine. Reasons for developing AKI, include dehydration, low blood pressure, medication and infection. When the kidneys stop working, there can be a build-up of toxins and fluid. It is extremely important to identify a patient's fluid status as too little can cause further damage to the kidneys and too much can be harmful. Assessment is varied and often inaccurate and there needs to be a standard approach to fluid assessment.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is the sudden and recent reduction in kidney function. This can be detected by measuring a rise in blood creatinine level or from a reduction in urine. Reasons for developing AKI, include dehydration, low blood pressure, medication and infection. When the kidneys stop working, there can be a build-up of toxins and fluid. It is extremely important to identify a patient's fluid status as too little can cause further damage to the kidneys and too much can be harmful. Assessment is varied and often inaccurate and there needs to be a standard approach to fluid assessment.

Aim:

To develop an Enhanced Fluid Assessment Tool for patients with AKI.

Workstream 1:

Aim: To identify what methods are useful to assess fluid in a patient with AKI. The fluid assessment techniques that are useful and are used, bioimpedance and patient reported signs and symptoms.

Workstream 2:

Aim: To identify the best methods of determining fluid status in a patient with AKI The findings from Workstream 1 will be used to rank the most useful fluid assessment techniques. This will lead to the development of the enhanced fluid assessment tool.

Workstream 3:

Aim: To assess if the tool is practical and clinically useful in determining a patient's fluid status.

The terminology and language will be reviewed and the tool will be used to assess patients and to determine the patients fluid status.

ELIGIBILITY:
Inclusion Criteria:

* Workstream 1 and 3 (phase 3):

Patients who will be included in the study will be Adult patients (over 18 years old) identified as having an acute kidney injury (AKI) within 72 hours of admission to hospital.

Workstream 2:

Experts in fluid assessment (Doctors, Nurses and AHPs). Persons included will be experts in their field of practice and have a recognised expertise in fluid assessment.

Workstream 3:

Phase 1: Experts in fluid assessment (Doctors, Nurses and AHPs). Phase 2: Staff nurses currently working on a clinical ward.

Exclusion Criteria:

* Patients who have kidney failure requiring dialysis or who are being conservatively managed.
* Patients who are receiving end of Life (EoL) care.
* Patients who have a pacemaker as this interferes with bioimpedance (WS1+3).
* There is no baseline creatinine.
* The patient has acquired an AKI 72 hours after admission to hospital.
* The patient has acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient admitted into hospital that has an acute kidney injury within the first 72 hours of admission.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
To identify the components of clinical assessment deemed useful in determining fluid status in patients with AKI. | Within 72 hours of admission
  Identifying the components of a volume assessment as defined in RCP (2015) Acute care toolkit and a scoping review on fluid assessment. Assessment includes; physiological parameters including blood pressure, weight changes, and physical examination, including identifying any signs of oedema or dehydration and history taking.

SECONDARY OUTCOMES:
To identify fluid status of patients with AKI using multiple assessments, including Bioimpedance, objective and subjective clinical assessments. | Within 72 hours of admission
  Bioimpedance measures fluid status and location of this fluid within the body.
To identify patient-focussed signs and symptoms of hydration in AKI | Within 72 hours of admission
  The patient with acute kidney injury will be asked to describe their signs and symptoms relating to acute kidney injury.
To evaluate whether fluid status of patients is related to: Stage of AKI, Cause of AKI, Length of stay, NEWS2 Measurements | At 30 days after admission
  To identify descriptive data from the patients medical notes.
To evaluate whether fluid status of patients is related to: Physical assessment (JVP, oedema, skin, respiratory, lying and standing BP, passive leg raise), Blood results: urea and creatinine, electrolytes, albumin, haemoglobin and bicarbonate. | Within 72 hours of admission
  Comparison between patients in different fluid status groups will be compared using t-tests (or non-parametric comparisons), or Chi squared (χ2) tests. Multi variable models will be explored to evaluate the relationship of measured variables to fluid status using logistic models.
To evaluate whether fluid status is related to: Fluid balance chart/ trends and documentation (positive or negative balance) , Weight trends, Charlson Co-morbidity index | At 30 days since admission
  A multivariate analysis of clinical characteristics (specifically as listed in the primary objective) to investigate their predictive effect for mortality at 30 days. Variables that are significant in univariate models at the 10% level will be then included in a multivariable regression analysis.
To evaluate whether fluid status is related to: Outcome: Renal Replacement therapy (RRT) during admission/ Recovery of kidney / dialysis dependence at 30 days/ Intensive care admission • Mortality (hospital 30-days) • Readmission (within 30 days) | At 30 days after admission
  A multivariate analysis of clinical characteristics (specifically as listed in the primary objective) to investigate their predictive effect for mortality at 30 days. Variables that are significant in univariate models at the 10% level will be then included in a multivariable regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Pattison, Principal Investigator — East and North Herts
Locations (1):
- East and North Hertfordshire NHS Trust, Lister Hospital, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: No